CLINICAL TRIAL: NCT04671563
Title: A Randomized, Single-Dose, Parallel-Group Study to Evaluate thePharmacokinetic Profiles of Two Formulations of Tenofovir Disoproxil Fumarate After Oral Administration in Healthy Volunteers Under Fasting Conditions
Brief Title: Pharmacokinetics of Two Formulation of Tenofovir Disoproxil Fumarate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yung Shin Pharm. Ind. Co., Ltd. (Industry)
Collaborators: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YSP-RKH3002-01
Record Dates: First submitted 2020-12-15; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Pharmacokinetic of Tenofovir in Healthy Subjects
MeSH Terms: interventions — Tenofovir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Viproof Film Coated Tablets 300mg (Experimental): Dosage form：Film-coated tablet Strength： 300 mg/tablet Dose：300 mg (one tablet, single oral dose)
  Interventions: Drug: Tenofovir Disoproxil Fumarate 300 MG
- Viread Tablets (Active Comparator): Dosage form：Film-coated tablet Strength： 300 mg/tablet Dose：300 mg (one tablet, single oral dose)
  Interventions: Drug: Tenofovir Disoproxil Fumarate 300 MG

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate 300 MG — One tablet of Viproof Film Coated Tablets or Viread Tablets will be orally administrated with 240 mL of water in the morning.

SUMMARY:
To evaluate pharmacokinetic profiles of Viproof Film Coated Tablets 300 mg manufactured by Yung Shin Parm. Ind. Co., Ltd., Taiwan and Viread Tablets manufactured by Patheon, Inc. in terms of plasma concentrations of tenofovir after a single oral dose of 300 mg tenofovir disoproxil fumarate in healthy subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female subjects between 20-45 years of age.
2. Body weight within 80-120% of ideal body weight.

   * Ideal body weight (kg) = [height (cm) - 80] *0.7 for male subjects
   * Ideal body weight (kg) = [height (cm) - 80] *0.6 for female subjects
3. Acceptable medical history and physical examination including:

   * no particular clinically significant abnormalities in electrocardiogram results within six months prior to dosing.
   * no particular clinical significance in general disease history within two months prior to dosing.
4. Acceptable biochemistry determinations (within normal limits or considered by the investigator or physician to be of no clinical significance) within two months prior to study drug dosing, which includes Serum Glutamic Oxaloacetic Transaminase (SGOT, same as AST), Serum Glutamic Pyruvic Transaminase (SGPT, same as ALT), Gamma-Glutamyl-Transpeptidase (γ-GT), alkaline phosphatase, total bilirubin, albumin, glucose, Blood Urea Nitrogen(BUN), uric acid, creatinine, total cholesterol and triglyceride (TG).
5. Acceptable hematology (within normal limits or considered by the investigator or physician to be of no clinical significance) within two months prior to study drug dosing, which includes hemoglobin, hematocrit, red blood cell count, white blood cell count with differentials and platelets.
6. Acceptable urinalysis (within normal limits or considered by the investigator or physician to be of no clinical significance) within two months prior to study drug dosing, which includes power of hydrogen (pH), blood, glucose, ketones, bilirubin and protein.
7. Females of childbearing potential practicing an acceptable method of birth control for the duration of the study.
8. Have signed the written informed consent to participate in the study.

Exclusion Criteria:

1. A clinically significant disorder involving the cardiovascular, respiratory, hepatic, renal, gastrointestinal, immunologic, hematologic, endocrine or neurologic system(s) or psychiatric disease (as determined by the investigator).
2. A clinically significant illness or surgery within four weeks prior to dosing (as determined by the investigator).
3. History of gastrointestinal obstruction, inflammatory bowel disease, gallbladder disease, pancreas disorder over last two years or history of gastrointestinal tract surgery over last five years.
4. History of kidney disease or urination problem over last two years deemed by the investigator to be clinically significant.
5. Known or suspected history of drug abuse within lifetime.
6. History of alcohol addiction or abuse within last five years as judged by the investigator.
7. History of allergic response(s) to tenofovir disoproxil fumarate or any other related drugs.
8. Evidence of chronic or acute infectious diseases.
9. Positive results for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), or human immunodeficiency virus (HIV).
10. Female subjects demonstrating a positive pregnancy screen prior to the study.
11. Female subjects who are currently breastfeeding.
12. Taking any drug known to induce or inhibit hepatic drug metabolism within four weeks prior to study drug dosing. Examples of inducers include: piperidines, carbamazepine, dexamethasone and rifampin. Examples of inhibitors include: cimetidine, diphenhydramine, fluvastatin, methadone and ranitidine.
13. Taking any prescription medications within four weeks or any nonprescription medications (excluding flu vaccination) within two weeks prior to study drug dosing.
14. Use of any investigational drug within four weeks prior to dosing.
15. Donating more than 250 mL of blood within two months prior to dosing or donating plasma (e.g. plasmapheresis) within two weeks prior to dosing.
16. Any other medical reason as determined by the investigator.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2020-05-09 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | Plasma sample: 0, 0.17, 0.33, 0.67, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48 and 72 hours post dose
  Area under the plasma concentration (AUC), peak concentration (Cmax), time to reach peak concentration (Tmax), elimination half-life (T1/2), total

SECONDARY OUTCOMES:
Adverse events and incidences | Within 1 hour before dosing, and 0.67, 12, 24, 36, 48 and 72 hours post dose

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan